CLINICAL TRIAL: NCT01466439
Title: Evaluation of Effect of Low and High-frequencies of Repetitive Transcranial Magnetic Stimulation (rTMS) by the Suppression of P50 Evoked Potential Component (rTMS-P50)
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) and P50 Evoked Potential Component
Acronym: rTMS-P50
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 09-181
Record Dates: First submitted 2011-10-19; First posted 2011-11-08 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Depression; Schizophrenia
Keywords: rTMS; P50; inhibitory; facilitatory; physiological process; brain changes
MeSH Terms: conditions — Depression; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high frequency rTMS (Other)
  Interventions: Procedure: high-frequency of repetitive transcranial magnetic stimulation (rTMS)
- low frequency rTMS (Other)
  Interventions: Procedure: low frequency of repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Procedure: high-frequency of repetitive transcranial magnetic stimulation (rTMS) — frequency of stimulation of 20 Hz
  Arms: high frequency rTMS
Procedure: low frequency of repetitive transcranial magnetic stimulation (rTMS) — frequency of stimulation of 1 Hz
  Arms: low frequency rTMS

SUMMARY:
The repetitive transcranial magnetic stimulation (rTMS) is a recent technique that has demonstrated its efficiency in both depression and schizophrenia. However if its efficiency has been recognized by the scientific community and the clinicians, its action on neurons and cerebral networks remains debated.

In the motor regions, the different rTMS studies generally use frequencies of stimulation of 1 to 40 Hz with differential effects; the low frequencies being associated with an inhibitory effect whereas highest frequencies have rather some facilitator effects as attested by the motor responses. What is valid for the motor system is not however necessarily applicable to other cerebral regions that have different neuronal organizations. If it is easy to observe these opposite effects of rTMS on the motor system (presence or absence of movements), these potential effects on more integrated cortex involved in high level functions have not been proved.

One of the possibilities to interpret the effects of the rTMS in no-motor cerebral regions would be to study the modifications of the EEG before and after rTMS and to see if a differential effect of the high and low frequencies of stimulation exists. Up to now, the studies having coupled these two techniques have observed modifications of the brain electric activity only during some seconds to minutes after rTMS, what appears in contrast with the clinical effects observed after a long delay (several days).

The contribution of our research resides in the use of the paradigm of suppression of P50 evoked potential component before and after rTMS tested with low and high frequencies of stimulation. This paradigm consists in two identical auditory stimuli presented at a very short interval (generally 500 milliseconds), the second sound generating a P50 wave of weaker amplitude than the first or being completely abolished in healthy subjects. However, this effect that has been well studied could result from an inhibitory action due to the gabaergic interneurons on the pyramidal neurons of the cortex. Thus, the investigators hypothesize that high frequency rTMS would have a facilitator effect on temporal lobe and so would induce no suppression of the P50 after-rTMS whereas low frequency rTMS would induce an inhibitory effect marked by a greater suppression of the P50.

Methods: 30 healthy subjects (of which 16 women) will be included after written consent. They will receive after randomization 2 sessions of rTMS in cross over at 1Hz and 20Hz at 30 days interval. An EEG and a P50 evoked potential will be done before and after rTMS. The site of stimulation will be determined by neuronavigation and will correspond to the maximal activation cluster generated by a language task during functional magnetic resonance imaging. The main judgment criterion is the S2/S1 ratio of the P50. The potential secondary effects will be evaluated (UKU adapted). The secondary criteria are the comparisons before and after rTMS of EEG spectrums in the alpha, beta and gamma bands.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects, right-handed, aged from 18 to 60 years
* written consent
* with social security

Exclusion Criteria:

* pregnancy, breastfeeding
* brain tumor or epilepsy
* psychiatric, neurological or ear-nose-throat disorders, current or past
* healthy subjects with psychotropic drugs or with substance abuses
* healthy subjects with tabacco weaning
* protected major with tutor
* counter-indication to MRI and rTMS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
P50 Ratio Stimulation 2/S stimulation 1 | day of stimulation (day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Pr Sonia Dollfus, MD, PhD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, department of psychiatry and explorations fonctionnelles neurologiques, Caen, France